CLINICAL TRIAL: NCT01609205
Title: Doppler Quantitative Evaluation and Follow-up Over 12 Months in RA Patients With Moderate and High Disease Activity Who Are Candidates for Biologic add-on Therapy With Adalimumab
Brief Title: Doppler Evaluation in RA Patients After Adalimumab.
Acronym: Muscara
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamed Rezaei (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Hamed Rezaei, Chief Arthritis, Inflammation department, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ClinTrid-US-1201; 2012-002573-62 (EudraCT Number)
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Adalimumab
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab 40 mg eow (totally 27 doses/patient) manufactured by Abbott will be distributed as add-on therapy to DMARD
  Other Names: Humira

SUMMARY:
The purpose is to study the relationship between RA disease activity based on Doppler quantification and the subsequent clinical response (EULAR response) to treatment with Adalimumab during 12 months. The purpose is also to compare the Doppler quantification with conventional clinical methods and semiquantitative Doppler assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years of age), male or female
* Rheumatoid arthritis according to the 1987 ACR or 2010 EULAR/ACR classification criteria
* Moderate to high disease activity
* Ongoing anti-rheumatic treatment with DMARD, with stable dosage during the last 3 months, and being a candidate for anti-TNF add-on therapy OR ongoing treatment with first anti-TNF therapy and being a candidate for switch to another anti-TNF therapy
* Women with child-bearing potential: use of an adequate method of contraception to avoid pregnancy throughout the study
* Signed Informed Consent *Signed Informed Consent must be obtained before any study specific procedures take place.

Exclusion Criteria:

* Biologic treatment with Adalimumab before inclusion
* Two or more ongoing biologic treatments before inclusion
* Treatment with other biologic treatment than anti-TNF therapy before inclusion
* Any contraindication for treatment with Adalimumab
* Intraarticular corticosteroid injection during the last 4 weeks before each follow-up visit
* Positive for tuberculosis or hepatitis B.
* Ongoing pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The proportion of different clinical (EULAR) response | 6 months from BL
  The primary endpoint will be the proportion of different clinical (EULAR) response (good, moderate, no response)* to add-on therapy with anti-TNF treatment at 6 months follow-up visit in patients with activity versus in those without activity measured by Doppler ultrasound at baseline.

SECONDARY OUTCOMES:
The proportion of patients with good response to add-on therapy | 6 and 12 months from BL
  The proportion of patients with good response to add-on therapy (measured by both Doppler and clinical assessment) at 6 and 12 months follow-up visits in two groups of patients, those who achieve low disease activity according to Doppler assessment at 3 months visit versus those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rydén Aulin, Phd, Study Chair — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Linköping University Hospital, Linköping
  - The karolinska Institute, Stockholm

IPD SHARING:
Plan to Share IPD: No